CLINICAL TRIAL: NCT04038541
Title: Prebiotic and Probiotic Treatment Trial in Multiple Sclerosis
Brief Title: Prebiotic vs Probiotic in Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Multiple Sclerosis Society (Other); Exegi Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AAAR9614
Record Dates: First submitted 2019-06-07; First posted 2019-07-31 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome (CIS)
Keywords: Prebiotics; Probiotics; Gut microbiome; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Prebiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: This is a randomized, interventional trial with a crossover design, in which participants will be taking either probiotic (commercially available Visbiome) or prebiotic (prebiotin prebiotic) for 6 weeks as the first agent. Then, participants enter a 6-week washout period. After the washout period, participants take the second agent for 6 weeks. After taking the second agent, participants again have a 6-week wash-out period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic/ Probiotic (Other): These subjects will be assigned to first receive prebiotics (Prebiotin Prebiotic Fiber Stick Pac) for 6 weeks. Then after a 6 week wash-out period, subjects will take probiotics (Visbiome®) for 6 weeks (followed again by a 6 week washout period).
  Interventions: Dietary Supplement: Prebiotics (Prebiotin Prebiotic Fiber Stick Pac); Dietary Supplement: Probiotics (Visbiome®)
- Probiotic/ Prebiotic (Other): These subjects will be assigned to first receive probiotics (Visbiome®) for 6 weeks. Then after a 6 week wash-out period, subjects will take (Prebiotin Prebiotic Fiber Stick) for 6 weeks (followed again by a 6 week washout period).
  Interventions: Dietary Supplement: Prebiotics (Prebiotin Prebiotic Fiber Stick Pac); Dietary Supplement: Probiotics (Visbiome®)

INTERVENTIONS:
Dietary Supplement: Prebiotics (Prebiotin Prebiotic Fiber Stick Pac) — Commercially available Prebiotin Prebiotic.
  2 packets (Inulin 4000 mg), Twice Daily (Total of 16 g Daily)
Dietary Supplement: Probiotics (Visbiome®) — Commercially available Probiotics Visbiome extra strength, which is a combination of live lactic acid bacteria probiotics that have been cultivated, freeze-dried and mixed in very high concentrations.
  2 packets (450 billion CFU), Twice Daily (Total of 3,600 billion Daily)

SUMMARY:
This is a randomized crossover-designed study to explore the immunologic effects of Prebiotics, as opposed to direct supplementation with beneficial bacteria (Probiotics) in the immune system of patients with MS and Clinically Isolated Syndrome (CIS). Eligible patients will take 6 weeks of two different supplements - Prebiotics and Probiotics. Participants will be randomly assigned to take either of two agents for 6 weeks as their first supplement. Then, participants enter a 6-week washout period. After the washout period, participants will take the second supplement for 6 weeks. After taking the second supplement, participants will have a 6-week washout period.

DETAILED DESCRIPTION:
Soluble fibers (prebiotics) are fermented by beneficial bacteria (probiotics) in the colon to produce short-chain fatty acids (SCFAs) which are the main source of nutrition for the cells in the gut. It has been reported that the fermentable fiber inulin and SCFAs may exert some beneficial effects including anti-inflammatory effect on the immune system. To date, the effect of supplementation with fermentable dietary fiber, such as prebiotics in patients with Multiple Sclerosis (MS) has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or older) diagnosed with MS (Relapsing-remitting type) or CIS and recruited within 10 years of symptom onset, and
* Adult patients receiving anti-CD20 therapy (rituximab or ocrelizumab) who have received at least one cycle at the time of recruitment

Exclusion Criteria:

* Active relapse within 3 months of enrollment
* Steroid use within 4 weeks of enrollment
* Antibiotics use within 3 months of enrollment
* Daily pre or prebiotic use within 3 months of enrollment
* Diagnosed with any of the autoimmune disorders: Rheumatoid Arthritis, Lupus, Celiac disease, Vitiligo, Psoriasis, Psoriatic Arthritis, Hashimoto's Thyroiditis, Graves' Disease, Sjogren's syndrome, Type 1 Diabetes, Scleroderma, Crohn's Disease, Ulcerative Colitis, Alopecia Areata.
* Had surgery of the GI tract in the last 5 years (with the exception of cholecystectomy and appendectomy)
* Had a major bowel resection
* Prior use of any of the following drugs: Mycophenolate/Cellcept, Cyclophosphamide/Cytoxan, Methotrexate/Novantrone, Azathioprine/Imuran, Cladribine/Leustatin/Mavenclad, Daclizumab/Zenepax, Alemtuzumab/Campath/Lemtrada
* Have any of the following active uncontrolled gastrointestinal (GI) illnesses:

  1. Crohn's disease, ulcerative colitis, indeterminate colitis
  2. Irritable bowel syndrome: moderate-severe
  3. Persistent or chronic diarrhea of unknown etiology
  4. Severe Chronic constipation or difficulties with defecation
  5. Persistent, infectious gastroenteritis, colitis or gastritis
  6. Clostridium difficile infection (recurrent)
  7. Gastric or intestinal ulcerations/GI bleeding
  8. Gastrointestinal or colonic malignancy: polyps, masses, dysplasia or cancer
* Active use of bismuth subsalicylate-containing products
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Peripheral Blood Mononuclear Cells (pBMCs) | Up to 24 weeks
  Measure the number of differentially expressed probe sets in the pBMCs post-supplementation, as compared to subject baseline. Probe sets will count as differentially expressed based on a threshold of pBH <0.05 and a Fold Change (FC) > ±2.
Change in Serum Neurofilament Light Concentration | Up to 24 weeks
  Change in serum neurofilament light concentration post-supplementation as compared to baseline. Serum neurofilament light (NfL) will be measured in terms of pg/ML.
Change in relative abundance of gut microbiome | Up to 24 weeks
  Changes in the gut microbiota in stool samples will be assessed as percent relative abundance at the genus level post supplementation as compared to baseline. Gut microbiota will be identified by extracting bacterial DNA from stool samples and performing metagenome shotgun sequencing.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale | Up to 24 weeks
  Modified Fatigue Impact Scale assesses fatigue effects in terms of physical, cognitive, and psychosocial functioning. The total core ranges from 0 - 20 (5 item version). Higher scores suggest a greater impact of fatigue on a patient's activities.
Bowel Control Scale | Up to 24 weeks
  Bowel Control Scale measures the impact of bowel control on lifestyle. The total score range from 0 - 26 (5 item version). Higher scores indicate greater bowel control issues.
Patient Determined Disease Steps | Up to 24 weeks
  Patient Determined Disease Steps assesses disability and walking ability in MS patients. Scores range from 0 (normal) to 8 (bedridden).
Multiple Sclerosis Rating Scale | Up to 24 weeks
  Multiple Sclerosis Rating Scale - Revised evaluates functional status to identify disability in domains other than walking. Scores range from 0 (normal status) to 4 (severe disability).
Patient Health Questionnaire | Up to 24 weeks
  Patient Health Questionnaire helps identify symptoms that could be related to depression. The total score ranges from 0 (None) to 27 (Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Farber, MD, Principal Investigator — Columbia University; Zongqi Xia, MD, Principal Investigator — University of Pittsburgh (Collaborator Site)
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - University of Pittsburg, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No